CLINICAL TRIAL: NCT05616403
Title: Textbook Outcome as a Composite Outcome Measure in Laparoscopic Pancreaticoduodenectomy: a Retrospective, Observational Study
Brief Title: Textbook Outcome as a Composite Outcome Measure in Laparoscopic Pancreaticoduodenectomy
Status: Completed | Type: Observational
Sponsor: Tongji Hospital (Other)
Collaborators: West China Hospital (Other); The Second Hospital of Hebei Medical University (Other); Hunan Provincial People's Hospital (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); Chinese PLA General Hospital (Other); Sir Run Run Shaw Hospital (Other); The Affiliated Hospital of Xuzhou Medical University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); First Affiliated Hospital of Chongqing Medical University (Other); Fujian Medical University Union Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Nanjing Medical University (Other); The First Hospital of Jilin University (Other); Zhejiang University (Other); Huadong Hospital (Other)
Responsible Party: Principal Investigator, Renyi Qin, Professor in Surgery, Chief Physician, Director of Surgical Supervision Department, Deputy Director of Institute of Hepatobiliary&Pancreatic, Director of Department of Biliary-Pancreatic Surgery, Tongji Hospital
Other Study IDs: TJDBPS13
Record Dates: First submitted 2022-11-08; First posted 2022-11-15 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Pancreatic Neoplasms
Keywords: textbook outcome; laparoscopic pancreaticoduodenectomy; composite outcome measure; hospital variation
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Textbook outcome group: Achieving textbook outcome after laparoscopic pancreaticoduodenectomy
  Interventions: Other: No intervention
- Non-Textbook outcome group: Not achieving textbook outcome after laparoscopic pancreaticoduodenectomy
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational study without any intervention

SUMMARY:
This is a multicenter, retrospective, observational study. Textbook outcome is a composite outcome measure for surgical quality assessment. The aim of this study was to assess textbook outcome following laparoscopic pancreaticoduodenectomy in China, identify factors independently associated with achieving textbook outcome and analyze hospital variations regarding the textbook outcome after case-mix adjustment.

DETAILED DESCRIPTION:
Laparoscopic pancreaticoduodenectomy (LPD) remains one of the most complex and technically challenging procedures in pancreatic surgery, although LPD has developed rapidly worldwide in recent years. Traditionally, quality assessment of LPD has mainly focused on individual outcome measures such as morbidity, mortality, operative time, operative blood transfusion, readmission rates and length of hospital stay. However, individual outcome parameters do not reflect the multiple facets of the whole surgical procedure and do not measure actual variations among different hospitals. In this context, several outcome experts have suggested that composite measures of surgical quality may be better than individual outcome parameters to compare hospital performance. Textbook outcome (TO) is such a composite outcome measure of multiple desirable outcome metrics, which was first proposed in 2013 by Dutch colorectal surgeons in order to give a comprehensive summary of hospital performance. TO is realized when all of the desired outcome parameters are achieved following surgery and represents the optimal ("textbook") hospitalization.

Although several studies on TO in pancreatic surgery have been reported, relevant data on LPD are lacking, especially from China. The objective of this study was to assess TO among patients undergoing LPD in China, identify factors independently associated with achieving TO and analyze hospital variations regarding the TO after case-mix adjustment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients underwent laparoscopic pancreaticoduodenectomy.
2. Aged 18 to 75 years old.

Exclusion Criteria:

1. Peritoneal seeding or metastasis to distant sites.
2. Incomplete clinical data

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients underwent laparoscopic pancreaticoduodenectomy from 16 high-volume pancreatic centers in China from January 2010 and August 2016.
Sampling Method: Non-Probability Sample
Enrollment: 1029 (Actual)
Dates: Start 2010-01-18 (Actual); Primary Completion 2016-08-28 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Textbook outcome | up to 90 days
  Textbook outcome was defined as the absence of postoperative pancreatic fistula, postpancreatectomy hemorrhage, bile leakage, severe complications (Clavien-Dindo grade ≥ Ⅲ), in-hospital or 30-day mortality, and readmission within 30 days after discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Renyi Qin, MD, Study Director — Department of Biliary-Pancreatic Surgery, Affiliated Tongji Hospital
Locations (1):
- Department of Biliary and Pancreatic Surgery, Tongji Hospital, Affiliated Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

REFERENCES:
- [Derived] Wu Y, Peng B, Liu J, Yin X, Tan Z, Liu R, Hong D, Zhao W, Wu H, Chen R, Li D, Huang H, Miao Y, Liu Y, Liang T, Wang W, Yuan J, Li S, Zhang H, Wang M, Qin R; Minimally Invasive Treatment Group in the Pancreatic DiseaseBranch of China's International Exchange and Promotion Association for Medicine and Healthcare (MITG-P-CPAM). Textbook outcome as a composite outcome measure in laparoscopic pancreaticoduodenectomy: a multicenter retrospective cohort study. Int J Surg. 2023 Mar 1;109(3):374-382. doi: 10.1097/JS9.0000000000000303. PMID 36912568